CLINICAL TRIAL: NCT05863429
Title: Observational Study to Evaluate the Effectiveness, Immunogenicity and Safety of Inactivated COVID-19 Vaccine (TURKOVAC) Application
Brief Title: Observational National Vaccine Study
Status: Completed | Type: Observational
Sponsor: Health Institutes of Turkey (Other Government)
Responsible Party: Sponsor
Other Study IDs: TBS-VAC-COV-TUR-GF4.07
Record Dates: First submitted 2023-02-10; First posted 2023-05-18 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: COVID-19 Infection
Keywords: COVID-19; Effectiveness; Immunogenicity; Safety; Observational
MeSH Terms: conditions — COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Blood samples from volunteers who accepted the study will be used to evaluate the long-term safety and immunogenicity of the TURKOVAC vaccine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Individuals who have never been vaccinated against COVID-19: Individuals who have never been vaccinated against COVID-19 and who have applied to the study centers to be vaccinated with TURKOVAC within the scope of the routine vaccination program.
  Interventions: Biological: Taking biological samples (blood) and keeping records with phone calls
- Previously primary vaccinated individuals: 1. Those who have previously received two doses of Sinovac - Coronavac vaccine, who will receive the booster vaccine for the first time as TURKOVAC;
  2. Those who have previously received two doses of the BioNTech Comirnaty vaccine, who will receive the booster vaccine for the first time as TURKOVAC;
  3. Those who have previously received the primary vaccination of Sinovac - Coronavac Vaccine and who have received at least one dose of the booster vaccine of TURKOVAC and have accepted the second booster dose vaccination,
  4. Individuals who have previously received the primary vaccination of the BioNTech Comirnaty Vaccine and who have received at least one dose of the booster vaccine of the TURKOVAC and who have agreed to the second booster dose vaccination.
  Interventions: Biological: Taking biological samples (blood) and keeping records with phone calls
- Individuals who have only received TURKOVAC vaccine before: Only individuals who have previously been vaccinated of TURKOVAC will also be invited to be included in the study retrospectively.
  Interventions: Biological: Taking biological samples (blood) and keeping records with phone calls

INTERVENTIONS:
Biological: Taking biological samples (blood) and keeping records with phone calls — Within the scope of the study, no intervention will be made to the participants. According to the vaccination program implemented in Turkey, subjects who apply to the study centers for TURKOVAC vaccine will be invited to the study.

SUMMARY:
To assess the long-term safety of TURKOVAC in individuals who have not previously received the COVID-19 vaccine or who have received their primary vaccination with inactivated or mRNA vaccine, or who have received their primary vaccination with similarly inactivated or mRNA vaccine and who subsequently received the first dose or second dose of booster vaccine, who meet the inclusion/exclusion criteria of the study.

DETAILED DESCRIPTION:
The primary objective of the study was to evaluate the long-term safety of TURKOVAC in individuals who had never received a COVID-19 vaccine before, or who received their primary vaccination with inactivated or mRNA vaccine, or who received their primary vaccination with similarly inactivated or mRNA vaccine, and who subsequently received a first dose or second dose of booster vaccine, in individuals who met the inclusion/exclusion criteria of the study. The secondary objective of the study was to evaluate the immunogenicity of TURKOVAC in individuals who meet the inclusion/exclusion criteria of the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who meet all of the following criteria will be included in the study:

  1. Individuals aged 18 and over,
  2. Individuals who have never had a COVID-19 vaccine before OR who have received COVID-19 mRNA or inactivated vaccines in the primary vaccination and have selected TURKOVAC as the booster dose (3rd dose and 4th dose),
  3. Individuals who have not had COVID-19 during the last trimester,
  4. Only for subjects who will receive 4th dose of vaccine: Those who have received the third dose of TURKOVAC vaccine and those who have spent at least 90 days since the third dose,
  5. Individuals who agree to provide blood samples and verifiable identification information (in accordance with local regulations), who may be contacted by the investigator during the study and who may come into contact with the investigator,
  6. Individuals who will be able to voluntarily understand and sign informed consent,
  7. Individuals who accept phone calls to be made to them for the purpose of collecting safety-related data.

Exclusion Criteria:

* Subjects who meet one of the following criteria will be excluded from the study.

  1. For subjects who will receive primary vaccination: Individuals who have received any vaccine and/or flu vaccine within 14 days prior to the COVID-19 vaccine.
  2. Individuals who have chosen a vaccine other than TURKOVAC as a booster dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults aged 18 years and older
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse reactions | 3 - 7 days after vaccination
  Incidence of adverse reactions in all subjects within 3 - 7 days after vaccination (phone call).
Incidence of Serious Adverse Events (SAE) | 365 days after vaccination
  Incidence of Serious Adverse Events (SAE) up to 365 days after vaccination in all subjects

SECONDARY OUTCOMES:
Neutralizing antibody (pseudo neutralization-Neutralizing Anti Spike/RBD Antibody) levels | Immediately before the first dose of TURKOVAC vaccine (day 0) and on the following days of 28 (±2 days), 48 (±5 days), 84 (±5 days), and 168 (±10 days)
  Neutralizing antibody (pseudo neutralization-Neutralizing Anti Spike/RBD Antibody) levels (from subjects available) immediately before the first dose of TURKOVAC vaccine (day 0) and on the following days of 28 (±2 days), 48 (±5 days), 84 (±5 days), and 168 (±10 days)

OTHER OUTCOMES:
Microneutralization levels | Immediately before the first dose of TURKOVAC vaccine (day 0) and on the following days 28 (±2 days), 48 (±5 days), 84 (±5 days), and 168 (±10 days)
  Microneutralization levels (from subjects available) immediately before the first dose of TURKOVAC vaccine (day 0) and on the following days 28 (±2 days), 48 (±5 days), 84 (±5 days), and 168 (±10 days)
Determine the confirmed COVID-19 case rates | At least 14 days after the second dose of TURKOVAC vaccine
  To determine the confirmed COVID-19 case rates by symptomatic RT-PCR at least 14 days after the second dose of TURKOVAC vaccine
Neutralizing antibody (pseudo neutralization-Neutralizing Anti Spike/RBD Antibody) levels and microneutralization levels | Before the fourth dose of TURKOVAC vaccine is given and on the 28th (±2 days) day following the booster dose of vaccine
  Neutralizing antibody (pseudo neutralization-Neutralizing Anti Spike/RBD Antibody) levels and microneutralization levels (from subjects available) just before the fourth dose of TURKOVAC vaccine is given and on the 28th (±2 days) day following the booster dose of vaccine

CONTACTS AND LOCATIONS:
Overall Officials: İhsan Ateş, Assoc. Prof., Study Director — Assoc. Prof.
Locations (8):
- Turkey (Türkiye) (8):
  - Ankara City Hospital Internal Medicine Clinic, Ankara
  - T.R. Ministry of Health Abant Izzet Baysal University Training and Research Hospital, Bolu
  - Eskişehir City Hospital Internal Medicine, Eskişehir
  - T.R. Ministry of Health Kartal Dr. Lütfi Kirdar City Hospital Infectious Diseases, Istanbul
  - Kayseri City Training and Research Hospital, Department of Infectious Diseases and Clinical Microbiology, Kayseri
  - Erciyes University Faculty of Medicine, Department of Infectious Diseases and Clinical Microbiology, Kayseri
  - Health Sciences University Derince Training and Research Hospital, Kocaeli
  - Health Sciences University Kanuni Training and Research Hospital Infectious Diseases and Clinical Microbiology, Trabzon